CLINICAL TRIAL: NCT06403020
Title: Ultrasound-guided Quadratus Lumborum Block Versus Rectus Sheath Block in Paraumbilical Hernia in Adults: A Prospective Randomized Study
Brief Title: Ultrasound-guided Quadratus Lumborum Block Versus Rectus Sheath Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, professor, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R321.
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Quadratus Lumborum Block and Rectus Sheath Block
Keywords: quadratus lumborum block; rectus sheath block
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: In this randomized double blinded study, patients will be allocated randomly into two groups by a computer generated sequence using closed envelope method. Group Q (n=23) will have qadratus lumboroum (QL) block.
  Group R (n=23) will have rectus sheath (RS) block.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Q (Active Comparator): Group Q (n=23) will have a qadratus lumboroum (QL) block.
  Interventions: Procedure: Block
- Group R (Active Comparator): Group R (n=23) will have a rectus sheath (RS) block.
  Interventions: Procedure: Block

INTERVENTIONS:
Procedure: Block — qadratus lumboroum (QL) block

SUMMARY:
In this study we will compare the effectiveness of quadratus lumborum block and rectus sheath block in postoperative pain management after paraumbilical hernia repair

DETAILED DESCRIPTION:
patients will be allocated randomly into two groups by a computer generated sequence using closed envelope method. Group Q (n=23) will have qadratus lumboroum (QL) block.

Group R (n=23) will have rectus sheath (RS) block. Surgery will be performed by the same surgeon and the block also will be done by same anesthesiologist who will not be involved in postoperative assessment.

All patients will have a preoperative history taking, clinical examination and routine preoperative laboratory investigations will be done. Patients also will be learned how to deal with the VAS score before surgery. The visual analog scale (VAS) is a pain score at which a 10-cm line with two ends "no pain" on the left end and the "worst pain" on the right end, used to track pain for a patient or to compare pain between patients.(12,13) At operating room (OR), patients will be monitored by noninvasive blood blood pressure(NABP), peripheral oxygen saturation (spo2) and and electrocardiogram ( ECG). A peripheral intravenous cannula will be inserted. Patients will be premedicated by midazolam (1-2 mg), and they will be pre oxygenated 3-5 minutes before induction of anesthesia. General anesthesia will be given using propofol 2-3mg/kg intravenous(IV), fentanyl 1-2µg/kg IV and atracurium 0.5 mg/kg IV as a muscle relaxant to facilitate intubation. Anesthesia will be maintained by isoflurane and atracurium 0.1-0.2 mg/kg every 20-30 minutes. Patients will be mechanically ventilated with 50% O2 and 50% air keeping end-tidal CO2 between 30 - 35 mmHg. Fentanyl bolus doses of 0.5-1 mcg/kg will be given according to the changes of hemodynamic variables more than 20% base line).

After the end of the surgery, and by the use of (Philips clear vue350, Philip Healthcare, Andover MAO1810, USA) ultrasound probe to perform the block according to the patient group.

Group Q: patients will receive qadratus lumborum block. The procedure will be performed under complete aseptic conditions, in the supine position, with slight elevation of the ipsilateral pelvis using a high frequency probe (5---10 MHz),connected to an ultrasound unit in transverse orientation. the probe will be positioned transversely at the anterosuperior iliac spine (ASIS) and it will be moved cranially to visualize the three muscle layers of the abdominal wall. After identifying the external oblique muscle, the probe will be moved posterolaterally to find its posterior border (hook sign) with the internal oblique muscle below it forming a roof above the quadratus lumborum muscle. By tilting the transducer down, the middle layer of the thoracolumbar fascia will be seen as a bright hyperechoic line. A 21-gauge Stimuplex® A 100-mm needle (B. Braun Melsungen AG, Germany) will be inserted in-plane in the anterolateral-to-posteromedial direction. After negative aspiration 0.2-0.4 ml/kg of bupivacaine 0.25% will be injected slowly on each side. Group R: patients will receive rectus sheath block. Under complete antiseptic condition,the rectus muscle will be identified using a high frequency linear probe with a transverse orientation placed across the abdomen above the level of the umbilicus. Starting with the midline, the linea alba and rectus muscle on either side will be identified. The rectus sheath will appear as hyperechoic fascial plane encircling the rectus abdominis muscle. Using an in-plane technique, the needle (100-mm needle ) will be passed through the rectus abdominal muscle to reach the plane between it and the posterior rectus sheath. After negative aspiration 0.2-0.4 ml/kg of bupivacaine 0.25% will be injected slowly on each side, local anaesthetic will be seen peeling the rectus muscle off the posterior rectus sheath.

At the end of surgery, all anesthetics will be stopped, reversal of muscle relaxants will be given, patients will be extubated when they will able to breath spontaneously with adequate tidal volume. Patients will be transferred to postanesthesia care unit (PACU). All patients will receive paracetamol 1gm/kg every 8 hours. All treating and outcome assessors staff will be blinded to the group allocation of the patients. At the recovery room, patients will assess their pain using VAS score, and they will be monitored for postoperative pain. Patients will be transferred to the ward and will leave the post anesthesia care unit (PACU) with Aldrete score more than 9. (14) patient with Vas score ≥4, will recieve a rescue dose of morphine 3-5 mg IV.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-60 years old,
* American Society of Anesthesiology (ASA) I, Ⅱ,
* both sexes who will have PUH surgical repair under general anesthesia.

Exclusion criteria:

* Known allergy to any of the drugs that will be used in the study.
* Coagulation disorders.
* Infection at the site of injection.
* Liver or kidney disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue score | The first 24 hours postoperative
  Postoperative pain

SECONDARY OUTCOMES:
Age | 1 year
  Demographic data

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan to share

REFERENCES:
- [Result] Karaarslan E, Topal A, Avci O, Tuncer Uzun S. Research on the efficacy of the rectus sheath block method. Agri. 2018 Oct;30(4):183-188. doi: 10.5505/agri.2018.86619. PMID 30403273
- [Result] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787